CLINICAL TRIAL: NCT03493464
Title: BR55 Contrast Enhanced Ultrasound (CEUS) in Characterization of Ovarian Lesions
Brief Title: BR55 in Characterization of Ovarian Lesions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision; expiration of available study agent due to long recruitment timeline.
Sponsor: Bracco Diagnostics, Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: BR55-108
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of sixty (60) subjects will be evaluated in the study. The first 10 subjects enrolled in the study will receive BR55 at a dose of 0.03 mL/kg. Assuming these first 10 subjects will show technically adequate images, subsequent subjects enrolled in the study will continue to receive 0.03 mL/kg dose of BR55; otherwise, subjects will be switched to a 0.05 mL/kg dose of BR55.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subjects will receive a single dose of BR55 at 0.03 mL/kg or 0.05 mL/kg.
  Interventions: Drug: BR55

INTERVENTIONS:
Drug: BR55 — A novel targeted ultrasound contrast agent

SUMMARY:
This is an exploratory phase II, single center, open label, prospective study of BR55 CEUS for characterization of ovarian lesions in subjects with suspected ovarian cancer.

DETAILED DESCRIPTION:
A total of sixty (60) subjects scheduled to undergo salpingo-oophorectomy within 30 days of BR55 CEUS examination will be enrolled to obtain approximately 30 subjects with benign ovarian lesions and 30 with malignant ovarian lesions based on the truth standard (TS).

The first 10 subjects will receive BR55 at a dose of 0.03 mL/kg. Assuming these first 10 subjects will show technically adequate images, subsequent subjects enrolled in the study will continue to receive 0.03 mL/kg dose of BR55; otherwise, subjects will be switched to a 0.05 mL/kg dose of BR55.

The final cancer diagnosis will be obtained for all subjects by histopathology.

ELIGIBILITY:
Inclusion Criteria: Enroll a subject if he/she meets the following inclusion criteria:

* Is at least 18 years of age;
* Has an ovarian lesion that is visible and assessable with trans-vaginal ultrasound;
* Is scheduled to undergo salpingo-oophorectomy for suspected ovarian cancer not earlier than 24 hours and not later than 30 days following BR55 administration;
* Provides written Informed Consent and is willing to comply with protocol requirements.

Exclusion Criteria: Exclude a subject if the subject does not fulfill the inclusion criteria, or if any of the following conditions are observed:

* Is a pregnant or lactating female. Exclude the possibility of pregnancy:

  * by testing on site at the institution (serum βHCG) within 24 hours prior to the start of investigational product administration,
  * by surgical history (e.g., tubal ligation or hysterectomy),
  * by post-menopausal status with a minimum 1 year without menses;
* Has undergone prior systemic therapy for ovarian cancer;
* Has history of concurrent malignancy;
* Has history of any clinically unstable cardiac condition including class III/IV congestive heart failure;
* Has had any severe cardiac rhythm disorders within 7 days prior to enrolment;
* Has severe pulmonary hypertension (pulmonary artery pressure >90mmHg) or uncontrolled systemic hypertension and/or respiratory distress syndrome;
* Has open and/or non-healing wounds in the chest, abdomen and pelvis;
* Has other systemic vascular abnormalities associated with neovascularization, such as macular degeneration, that in the opinion of the investigator could significantly affect the ability to evaluate the effects of BR55;
* Is participating in a clinical trial or has participated in another trial with an investigational compound within the past 30 days prior to enrolment;
* Has previously been enrolled in and completed this study;
* Has any known allergy to one or more of the ingredients of the Investigational Product or to any other contrast media;
* Is determined by the Investigator that the subject is clinically unsuitable for the study;
* Has had major surgery, including laparoscopic surgery, within 3 months prior to enrolment;
* Has history of surgery to the ovaries or pelvic inflammatory disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 14 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luigia Storto, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 subjects scheduled to undergo salpingo-oophorectomy within 30 days of BR55 contrast-enhanced ultrasound (CEUS) examination were to be enrolled to obtain approx. 30 subjects with benign ovarian lesions and 30 with malignant ovarian lesions based on the Truth Standard (TS; histopathology). This study was terminated early due to expiration of available BR55, therefore, only 14 of the 60 anticipated participants in the study were enrolled.
Pre-assignment Details: A subject was to be enrolled in the study if the following inclusion criteria were met: was at least 18 years old; had an ovarian lesion that was visible and assessable with trans-vaginal ultrasound; was scheduled to undergo salpingo-oophorectomy for suspected ovarian cancer not earlier than 24 hours and not later than 30 days following BR55 administration; and provided written Informed Consent and was willing to comply with protocol requirements.
Groups:
- Treatment: All subjects received a single dose of BR55 at 0.03 mL/kg in this study. No subject received a single dose of BR55 at 0.05 mL/kg.
  BR55: A novel targeted ultrasound contrast agent
Period: Overall Study
Arm/Group | Treatment
Started | 14
Completed | 13
Not Completed | 1
Not completed — Surgery not performed | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled and dosed in the study who provided demographic information.
Arm/Group | Treatment
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 55.4 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Exposure to Investigational Product [Mean (Standard Deviation); unit: Actual Volume Administered (mL)] — All subjects received a single dose of BR55 at 0.03 mL/kg in this study. No subject received a single dose of BR55 at 0.05 mL/kg.
  Actual Volume Administered (mL) | 2.16 (0.246)

OUTCOME MEASURES:

1. Primary Outcome: Visual Assessment of BR55 Enhancement
Description: BR55-enhanced images will be visually assessed using a 3-point scale (no enhancement=no focal targeted, stationary imaging signal was detectable; weak enhancement=weak focal targeted imaging signal was detectable and considered possibly stationary; strong enhancement=well-defined and strong focal targeted imaging signal was detectable and considered as definitely stationary).
Time Frame: 30 minutes post-dose on Day 1
Population: All participants enrolled and dosed in the study with BR55 enhancement assessed at 30 minutes post-dose timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 14
Participants
  No enhancement | 5
  Weak enhancement | 6
  Strong enhancement | 3

2. Primary Outcome: Adverse Events
Description: Number of participants who received the contrast agent and experienced an adverse event.
Time Frame: 2 days (day of and 24 hours after BR55 administration)
Population: All participants enrolled and dosed in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 14
Participants | 3

ADVERSE EVENTS:
Time Frame: Safety monitoring began at the time of signing Informed Consent and continued for 24 hours after BR55 administration, up to 3 days.
Description: Any untoward medical non-pre-existing symptom or medically significant laboratory or instrumental (e.g., electrocardiographic) abnormality, as well as worsening of pre-existing ones were considered to be an adverse event. All untoward medical occurrences, as well as the intensity (mild, moderate, severe), relationship (reasonable or no reasonable possibility)
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=14)
Headache (Nervous system disorders) | 3 (3)
Itchiness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT03493464/Prot_SAP_000.pdf